CLINICAL TRIAL: NCT00463359
Title: A Pilot Study of the Treatment of Facial Nodular and Nodulocystic Basal Cell Carcinoma With Double Curettage and Cautery Followed by Application of Imiquimod to the Base
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); Glasgow Western Infirmary (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WN07DE002; EudraCT No: 2007-001961-14
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Basal Cell Carcinoma
Keywords: basal cell carcinoma; curettage; Imiquimod; treatment
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Curettage; Cautery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Imiquimod cream
Procedure: curettage and cautery

SUMMARY:
The purpose of this study is to determine recurrence rates of nodular Basal Cell Carcinomas on the face removed with curettage and electrodessication (cautery) followed by application of Imiquimod cream to the base and further to achieve lower recurrence rates than after treatment with curettage and electrodessication alone.

DETAILED DESCRIPTION:
Basal Cell Carcinomas (BCC) are the commonest form of skin cancer in the white population. The face is where they most frequently occur and the nodular BCCs are the commonest type. Curettage and cautery/electrodessication (C&C) has been an established way of management of nodular BCCs for years, being a simple surgical procedure readily performed in outpatient clinics with good aesthetic results and high cure rates. The purpose of this study is to determine recurrence rates of nodular BCCs on the face removed with C&C followed by application of Imiquimod cream to the base and further to achieve lower recurrence rates than after treatment with C&C alone. Imiquimod is an immune response modifier with anti-tumour effects already licensed for the treatment of superficial BCCs in the UK.

ELIGIBILITY:
Inclusion Criteria:

* Well-defined primary, not previously treated nodulo-cystic BCC
* Size of the lesions: ≤ 1cm diameter
* Facial lesions
* Patient compliance competent
* Patient physically able to apply the treatment (cream)

Exclusion Criteria:

* Recurrent lesions
* Superficial, morphoeic or pigmented BCC
* Lesions close to vital structures; i.e. where C&C is not considered a standard treatment (eyelids, inner canthus, free borders)
* Lesions within 1 cm of the eyelids, nose, lips and hairline
* Immunosuppressed patients
* Women in childbearing age, pregnancy and breast-feeding
* Ages <50 or >90
* Patients compliance incompetent
* Patients physically incapable to apply the treatment (cream)
* Patients with Gorlin Syndrome (nevoid Basal Cell Carcinoma syndrome)

Ages: 49 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50

PRIMARY OUTCOMES:
Basal Cell Carcinoma recurrence rates in 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lorna MacKintosh, Specialist Registrar, Principal Investigator — Western Infirmary; Areti Makrygeorgou, Staff Grade Dr, Study Chair — Western Infirmary
Locations (1):
- Dermatology Department, Western Infirmary, Glasgow, Lanarkshire, United Kingdom